CLINICAL TRIAL: NCT05942066
Title: Feasibility Study Aiming at Pre-Analytical Standardization of Whole Blood Processing for Liquid Biopsy Applications
Status: Recruiting | Type: Observational
Sponsor: Tethis S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: TET-23-001
Record Dates: First submitted 2023-06-15; First posted 2023-07-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Whole Blood; Liquid Biopsy; Plasma; White Blood Cells; Pre-Analytical Standardization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy donors: Participants who are in good health and willing to provide a blood sample

SUMMARY:
The goal of this feasibility study is to evaluate a new sample preparator called See.d.

After blood processing the instrument will produce a set of slides and a tube of plasma. These outputs could be used in further analysis in liquid biopsy applications.

DETAILED DESCRIPTION:
This feasibility study aims at the evaluation of a new instrument called See.d , to be used in conjunction with its accessories, Smart Bio Surface (SBS) slides and reagents, for preparation of cytological samples (seeded on SBS slides) and plasma from fresh whole blood (within 4-6 hours from collection).

Blood samples will be collected from healthy volunteers and will be used to test See.d performances. Moreover the possibility of develop a new version of the instrument with increased processing capability and to develop and optimize analytical protocols for liquid biopsy applications will be evaluated as exploratory objectives.

The only study procedure will be the collection of a blood sample from each participants; during this study 200 participants will be enrolled.

For its feasibility nature, no formal statistics has been planned for this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing and able to give and sign a written informed consent
* Aged 18 or above

Exclusion Criteria:

* Ongoing infections requiring antibiotic or antiviral treatment
* Known hemostasis/coagulation disorder
* Known Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Blood samples to be used in this clinical study will be collected from healthy volunteers, already willing to become blood donors and, for this reason, already going to be subjected to a venipuncture and a blood draw to evaluate their eligibility to blood donation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
SBS slides stability | 1 day (at the blood draw)
  Evaluation of the area of adhered cell nuclei on SBS slides
Reagents stability | 1 day (at the blood draw)
  Evaluation of total adhered cell count on SBS slides
cfDNA quality control | 1 day (at the blood draw)
  Evaluation of the ratio between cfDNA and genomic contaminant DNA
Feasibility of staining on slides produced by See.d | 1 day (at the blood draw)
  Qualitative assessment of staining positivity
Feasibility of using See.d SBS slides for subsequent analysis | 1 day (at the blood draw)
  Recovery of mock-Circulating Tumor Cells (CTCs)
Feasibility of using See.d plasma for subsequent analysis | 1 day (at the blood draw)
  Recovery of spiked reference DNA

CONTACTS AND LOCATIONS:
Overall Officials: Luca Santoleri, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study without an individual participant data sharing plan

REFERENCES:
- [Background] Alix-Panabieres C, Pantel K. Liquid Biopsy: From Discovery to Clinical Application. Cancer Discov. 2021 Apr;11(4):858-873. doi: 10.1158/2159-8290.CD-20-1311. PMID 33811121
- [Background] Xie S, Wang Y, Gong Z, Li Y, Yang W, Liu G, Li J, Hu X, Wang Y, Tong Y, Yuan P, Si Y, Kang Y, Mao Y, Qi X, Liu Y, Ou J, Li Z, Pan X, Lv Z, Kaji K, Guo L, Lu R. Liquid Biopsy and Tissue Biopsy Comparison with Digital PCR and IHC/FISH for HER2 Amplification Detection in Breast Cancer Patients. J Cancer. 2022 Jan 1;13(3):744-751. doi: 10.7150/jca.66567. eCollection 2022. PMID 35154443
- [Background] Seale KN, Tkaczuk KHR. Circulating Biomarkers in Breast Cancer. Clin Breast Cancer. 2022 Apr;22(3):e319-e331. doi: 10.1016/j.clbc.2021.09.006. Epub 2021 Sep 22. PMID 34756687
- [Background] Hench IB, Hench J, Tolnay M. Liquid Biopsy in Clinical Management of Breast, Lung, and Colorectal Cancer. Front Med (Lausanne). 2018 Jan 30;5:9. doi: 10.3389/fmed.2018.00009. eCollection 2018. PMID 29441349
- [Background] Ho TH, Bissell MCS, Kerlikowske K, Hubbard RA, Sprague BL, Lee CI, Tice JA, Tosteson ANA, Miglioretti DL. Cumulative Probability of False-Positive Results After 10 Years of Screening With Digital Breast Tomosynthesis vs Digital Mammography. JAMA Netw Open. 2022 Mar 1;5(3):e222440. doi: 10.1001/jamanetworkopen.2022.2440. PMID 35333365
- [Background] Hofvind S, Ponti A, Patnick J, Ascunce N, Njor S, Broeders M, Giordano L, Frigerio A, Tornberg S; EUNICE Project and Euroscreen Working Groups; Van Hal G, Martens P, Majek O, Danes J, von Euler-Chelpin M, Aasmaa A, Anttila A, Becker N, Pentek Z, Budai A, Madai S, Fitzpatrick P, Mooney T, Zappa M, Ventura L, Scharpantgen A, Hofvind S, Seroczynski P, Morais A, Rodrigues V, Bento MJ, Gomes de Carvalho J, Natal C, Prieto M, Sanchez-Contador Escudero C, Zubizarreta Alberti R, Fernandez Llanes SB, Ascunce N, Ederra Sanza M, Sarriugarte Irigoien G, Salas Trejo D, Ibanez Cabanell J, Wiege M, Ohlsson G, Tornberg S, Korzeniewska M, de Wolf C, Fracheboud J, Patnick J, Lancucki L, Ducarroz S, Suonio E. False-positive results in mammographic screening for breast cancer in Europe: a literature review and survey of service screening programmes. J Med Screen. 2012;19 Suppl 1:57-66. doi: 10.1258/jms.2012.012083. PMID 22972811
- [Background] Durand MA, Friedewald SM, Plecha DM, Copit DS, Barke LD, Rose SL, Hayes MK, Greer LN, Dabbous FM, Conant EF. False-Negative Rates of Breast Cancer Screening with and without Digital Breast Tomosynthesis. Radiology. 2021 Feb;298(2):296-305. doi: 10.1148/radiol.2020202858. Epub 2020 Dec 1. PMID 33258744
- [Background] Alavi N, Khan SH, Saadia A, Naeem T. Challenges in Preanalytical Phase of Laboratory Medicine: Rate of Blood Sample Nonconformity in a Tertiary Care Hospital. EJIFCC. 2020 Mar 20;31(1):21-27. eCollection 2020 Mar. PMID 32256286
- [Background] Carbone R, Marangi I, Zanardi A, Giorgetti L, Chierici E, Berlanda G, Podesta A, Fiorentini F, Bongiorno G, Piseri P, Pelicci PG, Milani P. Biocompatibility of cluster-assembled nanostructured TiO2 with primary and cancer cells. Biomaterials. 2006 Jun;27(17):3221-9. doi: 10.1016/j.biomaterials.2006.01.056. Epub 2006 Feb 28. PMID 16504283
- [Background] Zanardi A, Bandiera D, Bertolini F, Corsini CA, Gregato G, Milani P, Barborini E, Carbone R. Miniaturized FISH for screening of onco-hematological malignancies. Biotechniques. 2010 Jul;49(1):497-504. doi: 10.2144/000113445. PMID 20615202